CLINICAL TRIAL: NCT00227214
Title: Prevalence of Pneumococcal Meningitis in the Paediatric Population in Spain Four Years After the Marketing of Prevenar.
Brief Title: Study Evaluating Pneumococcal Meningitis in the Paediatric Population in Spain Four Years After the Marketing of Prevenar.
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Other Study IDs: 0887X-101539
Record Dates: First submitted 2005-09-12; First posted 2005-09-27 (Estimated); Last update posted 2010-06-28 (Estimated); Status verified 2010-06

CONDITIONS: Pneumococcal Meningitis
MeSH Terms: conditions — Meningitis, Pneumococcal

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The aim of this study is to determine the prevalence of pneumococcal meningitis in the paediatric population in Spain four years after the marketing of Prevenar. Also secondary objectives are: 1) to determine the clinical characteristics and outcome of the disease; and 2) to determine serotypes and antibiotic resistance patterns.

ELIGIBILITY:
Inclusion Criteria:

* All children from 0 up to 14 years with diagnosis of confirmed or probable pneumococcal meningitis or with diagnosis of suspected bacterial meningitis without bacterial or viral isolation will be included into the study.

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children from 0 up to 14 years of age with a diagnosis of confirmed or probable pneumococcal meningitis or with a diagnosis of suspected bacterial meningitis without bacterial or viral isolation.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2004-01; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (39):
- Spain (39):
  - A Coruña
  - Alcalá de Henares
  - Alcorcón
  - Arrasate / Mondragón
  - Badalona
  - Barakaldo
  - Barcelona
  - Barco de Valdeorras
  - Bilbao
  - Boadilla del Monte
  - Cee
  - El Escorial
  - Esplugues de Llobregat
  - Estella-Lizarra
  - Ferrol
  - Figueres
  - Getafe
  - Girona
  - Granollers
  - Leganés
  - Lleida
  - Lugo
  - Madrid
  - Monforte de Lemos
  - Móstoles
  - Ourense
  - Pamplona
  - Pontevedra
  - Reus
  - Ribeira
  - Sabadell
  - San Sebastián
  - Tarragona
  - Terrassa
  - Tudela
  - Verín
  - Vigo
  - Vitoria-Gasteiz
  - Zumarraga